CLINICAL TRIAL: NCT02566785
Title: Balance Activities and Strengthening to Improve Condition [BASIC]: Training for Elders With Heart Failure
Brief Title: Balance Training for Elders With Heart Failure
Acronym: BASIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: American Nurses Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0677-15-FB
Record Dates: First submitted 2015-09-28; First posted 2015-10-02 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Experimental): Those allocated to the intervention group will participate in a supervised group session exercise one time per week and be asked to exercise two more times per week at home.
  Interventions: Other: Balance Intervention
- Wait List Control Group (Other): The wait list control group will not participate in the intervention and will be asked to continue their usual activity level during the first 12 weeks and will receive the multi-component balance intervention during weeks 12-24.
  Interventions: Other: Balance Intervention

INTERVENTIONS:
Other: Balance Intervention — The multi-component balance intervention will be 1x per week in supervised group sessions and 2x a week sessions at home. Sessions will begin with a 5 minute warm up of major muscle groups using flexibility exercises and end with a cool down. Sessions will focus on improving static balance in the initial stages, then progress to dynamic balance.

SUMMARY:
Falls are the leading cause of injury-related deaths in older (≥ 65 y/) community dwelling heart failure (HF) patients. Fall risks are even greater for those with HF due to decreased exercise capacity, loss of skeletal muscle & medication side effects. Though resistance training (RT) is effective for improving skeletal muscle, it has only a modest effect on improving balance, which is comprised of peripheral sensory input central integration, & motor output. A multi-component intervention focusing on balance retraining & strengthening the muscles supporting static/dynamic balance & functional mobility is necessary.

This pilot study will evaluate the effect of a multi-component balance & RT intervention on physical function, balance, & falls in older (≥ 65 y/) community dwelling heart failure (HF) patients. The study will also explore perceptions related to outcomes & the intervention through focus groups, generate data on adherence and generate data on feasibility of conducting the BASIC Training intervention. The results of this study will be used to develop a targeted intervention to induce changes in elderly HF patients to prevent future falls; thus reducing costs, physical & emotional burdens related to falls; & effect a major difference in the quality of life.

The study will be once per week supervised group sessions & twice a week home sessions, and include 30 Second Sit-to-Stand, Modified Clinical Test of Sensory Interaction on Balance, Activity Specific Balance Confidence Scale, Timed Up & Go, Dynamic Gait Index.

DETAILED DESCRIPTION:
Purpose: The purpose of this pilot study is to evaluate the effect of a multi-component balance and resistance training [RT] intervention on physical function, balance, and falls in older [≥ 65 y/o] community dwelling heart failure [HF] patients. The study aims: 1] Pilot test multi-component balance activities and RT intervention on primary outcomes. 2] Explore perceptions related to outcomes and the intervention through focus groups. 3] Generate pilot data on adherence. 4] Generate pilot data on feasibility of conducting the BASIC Training intervention.

Background/Significance: Falls are the leading cause of injury-related deaths in this age group. Fall risks are even greater for those with HF due to decreased exercise capacity, loss of skeletal muscle and medication side effects. Though RT is effective for improving skeletal muscle, it has only a modest effect on improving balance, which is comprised of peripheral sensory input central integration, and motor output. A multi-component intervention focusing on balance retraining and strengthening the muscles supporting static/dynamic balance and functional mobility is necessary.

Methods: Design - Randomized, two-group with wait list control, repeated measures experimental design. Sample/ Setting - 40-50 participants recruited from a medical center heart failure clinic; supervised group sessions conducted in the center's health and wellness center. Procedures - Participants will be randomized to the intervention group or the wait list control group. Focus groups pre/post intervention. The intervention will be administered in 1x per week supervised group sessions and 2x a week home sessions. Instruments - 30 Second Sit-to-Stand, Modified Clinical Test of Sensory Interaction on Balance, Activity Specific Balance Confidence Scale, Timed Up and Go, Dynamic Gait Index.

Analysis Plan: Aim 1- independent t-test to compare change scores from baseline to the end of the first 12 week period for the intervention group with the wait list control group. A second analysis will combine data from the delayed intervention period for the wait list control group with that from the first 12 week period for the intervention group to test change. Supplemental analysis, involving only data from intervention group, will test whether change is sustained at 24 weeks. Aim 2 - thematic analysis conducted with focus group data. Aim 3 - adherence assessed by group session attendance and home activities completed. Aim 4 - assess and report logistics of conducting the study.

Nursing Relevance/Implications: This pilot study will initiate the process of developing a targeted intervention to induce changes in elderly HF patients to prevent future falls; thus reducing costs, physical and emotional burdens related to falls; and effect a major difference in the quality of life for this population.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or greater;
* New York Heart Association class II and III,
* community dwelling;
* able to speak and read English,
* must have written permission from cardiologist to participate.

Exclusion Criteria:

* wheel chair dependency;
* history of significant residual neurologic deficits [e.g.: recent stroke];
* recent history of whiplash or concurrent complaints of neck pain;
* recent fracture or lower extremity surgery. Participants will be screened for cognitive dysfunction and must pass the Mini-Mental State Examination [with a score at or above 23 points].

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2016-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita L McGuire, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, College of Nursing, Lincoln, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2015 through June 2016 at the Heart Failure Improvement Program of a regional hospital.
Period: Overall Study
Arm/Group | Intervention Group | Wait List Control Group
Started | 15 | 18
Completed | 14 | 15
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Worsening condition | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Wait List Control Group | Total
Number analyzed (Participants) | 15 | 18 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 15 | 18 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 7 | 10 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 18 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Pre/Post Scores on the 30 Second Sit to Stand Test Will be Used to Detect Any Changes in Leg Strength and Endurance That Occur During the 12 Week Group Exercise Sessions.
Time Frame: Baseline and 12 weeks
Population: Two of the participants in the WLC group were there for testing at 12 weeks.
Measure: Mean (Standard Deviation); unit: number of sit to stand cycles
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 14 | 13
number of sit to stand cycles
  Baseline | 6.9 (4.2) | 6.5 (3.6)
  12 Weeks | 7.9 (4.5) | 7.7 (5.4)

2. Primary Outcome: Dynamic Gait Index
Description: 8 increasingly challenging walking tasks (normal gait speed, changes in gait speed, walking with horizontal and vertical head movements, walking with pivot turn, walking over and around obstacles and stair climbing). A walkway path measured at 20 feet was used. A research assistance observed and scored all participants using a 0-3 scale, 0 = severe gait impairment, 1 = moderate gait impairment, 2 = mild/minimal impairment, 3 = normal gait, with a total possible scale range of 0 to 24 points. Scores ≤ 19 points was used to classify falling risk (Shumway-Cook et al. 1997).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 14 | 15
units on a scale
  Baseline | 18.9 (3.8) | 19.1 (4.6)
  12 Weeks | 20.9 (1.8) | 18.9 (4.4)

3. Secondary Outcome: Activity Balance Confidence Scale
Description: Total range = 0-100% Higher values represent better outcome Total score is averaged = total%/16 responses
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Group | Wait List Control Group
Number analyzed (Participants) | 14 | 15
units on a scale
  Baseline | 74.9 (17.3) | 74.1 (12.6)
  12 weeks | 72.1 (13.3) | 71.2 (15.8)

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Intervention Group | Wait List Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/18
Other Adverse Events (participants affected / at risk) | 1/15 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=15) | Wait List Control Group (N=18)
Fall from chair to knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fell from seated on chair to knees when attempting to stand during testing. Lowered gently to floor by balance team member who had a gait belt on participant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No